CLINICAL TRIAL: NCT04205370
Title: Sleep Behaviors in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Research Associate Professor, Neurology, Research Associate Professor, Obstetrics and Gynecology, Medical School and Associate Research Scientist, Dentistry, Department of Oral and Maxillofacial Surgery, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00140170
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sleep; Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Deactivated device (Active Comparator): Wear deactivated pregnancy coach device for the remainder of pregnancy.
  Interventions: Device: Deactivated Pregnancy Coach
- Active device (Experimental): Wear active device for remainder of pregnancy (including 3 day run-in period)
  Interventions: Device: Active Pregnancy Coach

INTERVENTIONS:
Device: Deactivated Pregnancy Coach — Naturalistic monitoring of their typical sleep patterns and behaviors
  Arms: Deactivated device
Device: Active Pregnancy Coach — The Pregnancy Coach will begin to deliver alerts when supine sleep is detected. Sleep metrics will be visible on the smartphone app.
  Arms: Active device

SUMMARY:
The researchers would like to know how long pregnant women spend in different positions during the night - and how often women change positions - across pregnancy. The researchers also want to see if the sleep monitor is able to improve sleep behaviors

ELIGIBILITY:
Inclusion Criteria:

* At least 28 weeks pregnant
* Receiving pre-natal care at Michigan Medicine
* Have either and Android or iPhone smartphone

Exclusion Criteria:

* Less then 28 weeks pregnant
* Receiving pre-natal care external to Michigan Medicine
* Does not poses a smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of sleep time spent in the supine position as measured by the Pregnancy Coach | Until delivery, approximately 12 weeks
  Will be conducted using the naturalistic arm (deactivated device). Simple descriptive statistics to report the average number of minutes and the average proportion of supine sleep per week.

SECONDARY OUTCOMES:
Proportion of sleep time spent with objective snoring as indicated by the Pregnancy Coach | Until delivery, approximately 12 weeks
  Will be conducted using the naturalistic arm (deactivated device). Proportion of time will be determined during each gestational week.
Proportion of participants where their 'going to sleep' position was the same as their dominant sleep position | Until delivery, approximately 12 weeks
  Will be conducted using the naturalistic arm (deactivated device). We will determine whether the "going to sleep" position during each gestational week is predictive of the most dominant sleep position.
Percentage of sleep position changes following alert from Pregnancy Coach | Until delivery, approximately 12 weeks
  Will be conducted using the intervention arm (active device). Percentage of sleep position changes in response to an alert from the Pregnancy Coach will be reported for each gestational week.

CONTACTS AND LOCATIONS:
Overall Officials: Louise O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not have plans to actively share data, however, they are open to collaboration following contact with the investigator.